CLINICAL TRIAL: NCT00930527
Title: Randomized Phase II Study of Omega-3-Fatty Acid on Joint Symptoms Induced by Aromatase Inhibitors in Breast Cancer Patients
Brief Title: Omega-3-Fatty Acid on Joint Symptoms Inducted by Aromatase Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed by sponsor.
Sponsor: Columbia University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Dawn L. Hershman, Associate Professor of Medicine & Epidemiology, Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAD8300
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid — 4g per day for 3 weeks
  Other Names: Lovaza

SUMMARY:
There are no data regarding the use of supplements to alleviate the musculoskeletal pain and stiffness inducted by the use of aromatase inhibitors. This study is designated to test the safety and efficacy of omega 3 fatty acid supplementation to alleviate musculoskeletal pain in postmenopausal breast cancer patients.

DETAILED DESCRIPTION:
There are no data regarding the use of these supplements in other types of musculoskeletal pain and discomfort, namely AI induced joint pain and joint stiffness. Given the lack of effective treatments for AI induced joint pain/ stiffness and the safety and efficacy of omega 3 fatty acid for musculoskeletal pain, it is therefore reasonable to test the efficacy of these dietary supplements in a population of postmenopausal breast cancer patients who experience joint pain related to aromatase inhibitors. Since women with hormone receptor positive breast cancer require long term hormonal therapy, an important objective is minimizing long term side effects to enhance patient compliance and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years
* Postmenopausal status defined as cessation of menses for >1 year or FSH >20 mIU/mL or bilateral oophorectomy.
* History of stage I, II or III hormone receptor-positive breast cancer, without metastatic disease
* Currently taking a third-generation aromatase inhibitor for at least 3 months
* Clinical symptoms of knee and/or hand joint pain and/or stiffness for at least 3 months prior to study entry
* Ongoing musculoskeletal pain/stiffness in hand and/or knee joints (50 or higher on the 100 point global assessment VAS) that started or increased since initiating aromatase inhibitor therapy, and has been present for at least 3 months.
* Patients must agree to refrain from use of omega-3-fatty acid from sources outside of this study
* If taking bisphosphonates, on a stable dose for at least 1 month and tolerating the dose. Patients must agree to refrain from initiating bisphosphonate use during the course of the study, therefore it is recommended that routine bone density testing be performed prior to enrollment or after completing trial.
* ECOG performance status 0-2.
* Signed informed consent

Exclusion Criteria:

* Use of omega-3-fatty acid within the past three (3) months
* Concurrent medical/arthritic disease that could confound or interfere with evaluation of pain or efficacy including: Inflammatory arthritis (e.g., rheumatoid arthritis, systemic lupus, spondyloarthropathy, psoriatic arthritis, polymyalgia rheumatica), gout, episodes of acute monarticular arthritis clinically consistent with pseudogout, Paget's disease affecting the study joint, a history of septic arthritis or avascular necrosis or intra-articular fracture of the study joint, Wilson's disease, hemochromatosis, alkaptonuria, or primary osteochondromatosis.
* History of significant collateral ligament, anterior cruciate ligament or meniscal injury of the index joint requiring surgery or non-weight bearing (requiring use of crutches or cane) for more than 3 weeks (minor ligamentous injury prior to 6 months is not an exclusion).
* History of bone fracture or surgery of the afflicted knees and/or hands within 6 months prior to study entry.
* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient.
* Allergy to, or history of significant clinical or laboratory adverse experience associated with omega-3 fatty acid
* Inability to understand and complete study questionnaires including questions requiring a visual analog scale (VAS) response.
* Inability to understand the study procedures and/or give written informed consent.
* Alcohol use in excess of 3 mixed drinks/day.
* Corticosteroid treatment as follows:

  1. Use of oral corticosteroids within the previous four weeks.
  2. Exposure to intramuscular corticosteroids within one month prior to entering the study.
  3. Administration of intra-articular steroids to the study joint, within 3 months of Randomization Visit.
  4. Administration of intra-articular steroids to any other joint, within 3 months of Randomization Visit.
* Intra-articular injection of hyaluronic acid or congeners into the study joint within 12 months.
* Topical analgesics (e.g., capsaicin preparations) to the study joint, or any oral analgesics (e.g., opiates, tramadol; with the exception of ibuprofen and acetaminophen) within 2 weeks of Randomization Visit or during the study.
* Implementation of any other medical therapy for arthritis within one month prior to entry.
* Other medications, unrelated to the patient's joint pain/stiffness must have been used at a stable dosage for at least 1 month. In addition, it should be anticipated that the dose of the concomitant medication will be stable during the entire treatment period.
* Participation in another clinical study with an investigational agent within the last 4 weeks.
* Exposure to omega-3-fatty acid within 3 months of Baseline Visit.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
A change in serum free and total estradiol levels. | At week 3

SECONDARY OUTCOMES:
A change in the frequency of analgesics consumed | At 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States